CLINICAL TRIAL: NCT02174172
Title: A Phase Ib Study of The Safety And Pharmacology of Atezolizumab (Anti-Pd-L1 Antibody) Administered With Ipilimumab, Interferon-Alpha, or Other Immune-Modulating Therapies in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study to Assess the Safety and Tolerability of Atezolizumab in Combination With Other Immune-Modulating Therapies in Participants With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO29322; 2014-000812-33 (EudraCT Number)
Record Dates: First submitted 2014-06-19; First posted 2014-06-25 (Estimated); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Solid Cancers
MeSH Terms: interventions — atezolizumab; Bevacizumab; Interferon alpha-2; Ipilimumab; obinutuzumab; peginterferon alfa-2a

ARMS (5):
- Arm A: Atezolizumab with Ipilimumab (Experimental): Participants will receive atezolizumab along with ipilimumab.
  Interventions: Drug: Atezolizumab; Drug: Ipilimumab
- Arm B: Atezolizumab with Interferon alfa-2b (Experimental): Participants will receive atezolizumab along with Interferon alfa-2b.
  Interventions: Drug: Atezolizumab; Drug: Interferon alfa-2b
- Arm C: Atezolizumab with PEG- interferon alfa-2a (Experimental): Participants will receive atezolizumab along with PEG- interferon alfa-2a.
  Interventions: Drug: Atezolizumab; Drug: PEG-interferon alfa-2a
- Arm D:Atezolizumab with PEG-interferon alfa-2a and Bevacizumab (Experimental): Participants will receive atezolizumab along with PEG- interferon alfa-2a and bevacizumab.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Drug: PEG-interferon alfa-2a
- Arm E: Atezolizumab with Obinutuzumab (Experimental): Participants will receive atezolizumab along with obinutuzumab or atezolizumab alone.
  Interventions: Drug: Atezolizumab; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Atezolizumab — Participant will receive atezolizumab 600 milligrams (mg) or 1200 mg by IV infusion q3w.
  Other Names: Tecentriq, RO5541267, MPDL3280A
Drug: Bevacizumab — Participant will receive Bevacizumab 15 milligrams per kilograms (mg/kg) IV infusion q3w.
  Other Names: Avastin®
  Arms: Arm D:Atezolizumab with PEG-interferon alfa-2a and Bevacizumab
Drug: Interferon alfa-2b — Participants will receive Interferon alfa-2b 3, 5, or 10 million international units subcutaneously every other day for up to 3 doses per week.
  Arms: Arm B: Atezolizumab with Interferon alfa-2b
Drug: Ipilimumab — Participants will receive Ipilimumab 1, or 3 mg/kg IV, single dose, or multiple-dose regimen q3w for up to 4 cycles (Cycle = 21 days).
  Arms: Arm A: Atezolizumab with Ipilimumab
Drug: Obinutuzumab — Obinutuzumab 1000 milligrams will be administered as pre-treatment on 2 consecutive days (Day -13 and Day -12) prior to treatment start with atezolizumab on Cycle 1, Day 1 (cycle length=21 days). An additional two doses of obinutuzumab will be administered on Days 85 and 86 of study treatment (Cycle 5, Day 1 and Cycle 5, Day 2).
  Arms: Arm E: Atezolizumab with Obinutuzumab
Drug: PEG-interferon alfa-2a — Participant will receive PEG-interferon alfa-2a 180 micrograms subcutaneous injection q3w for a total of 6 cycles (Cycle = 21 days).
  Other Names: Pegasys®
  Arms: Arm C: Atezolizumab with PEG- interferon alfa-2a; Arm D:Atezolizumab with PEG-interferon alfa-2a and Bevacizumab

SUMMARY:
This global, multicenter, open-label study will evaluate the safety and tolerability of atezolizumab in combination with other immune-modulating therapies in the treatment of selected advanced or metastatic malignancies. The atezolizumab plus ipilimumab arm (Arm A) will focus primarily on participants with advanced or metastatic non-small cell lung cancer (NSCLC). The atezolizumab plus interferon alfa-2b arm (Arm B), plus pegylated interferon alfa-2a (PEG-interferon alfa-2a, Arm C), and atezolizumab plus PEG-interferon Alfa-2a plus bevacizumab (Arm D) will enroll participants with advanced or metastatic renal cell carcinoma (RCC), metastatic NSCLC and melanoma. The atezolizumab plus obinutuzumab) (Arm E) will enroll participants with recurrent and/or metastatic (R/M) head and neck squamous cell carcinoma (HNSCC). Atezolizumab will be administered as intravenous (IV) infusion every 3 weeks (q3w).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented locally advanced or metastatic solid tumors meeting the following study drug-specific criteria:
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Life expectancy greater than or equal to (>/=) 12 weeks
* Measurable disease, as defined by RECIST v1.1
* Adequate hematologic and end organ function as confirmed by laboratory results within 14 days prior to the first study treatment

Inclusion criteria specific to Arm A: Atezolizumab+ Ipilimumab

* Escalation stage: NSCLC participants
* Mandatory biopsy cohort: NSCLC or melanoma atezolizumab
* Prior atezolizumab-treated cohort: participants with NSCLC or melanoma previously treated with atezolizumab

Inclusion criteria specific to Arm B: Atezolizumab+ Interferon alfa-2b

* Escalation stage: RCC or melanoma participants
* Expansion stage: RCC or melanoma participants
* Mandatory biopsy cohort: RCC or melanoma participants
* Prior immunotherapy-treated cohort: participants with RCC, NSCLC, or melanoma previously treated with programmed death-ligand 1 (PD-L1)/ Programmed death 1 (PD-1)

Inclusion Criteria Specific to Arm C (Atezolizumab plus PEG-Interferon Alafa-2a):

- Cohort 1: participants with RCC

Inclusion Criteria Specific to Arm D (Atezolizumab plus PEG-Interferon Alfa-2a +Bevacizumab)

* Cohort 1: participants with metastatic RCC with no prior line of systemic therapy for metastatic disease
* Cohorts 2-3: disease progression during or after at least one previous systemic, anti-cancer treatment for locally advanced or metastatic non-squamous solid tumors; participants with sensitizing epidermal growth factor receptor (EGFR) mutations or anaplastic lymphoma kinase (ALK) rearrangements must have failed or are intolerant to prior treatment with EGFR or ALK inhibitors; participants with melanoma with actionable BRAF mutations (e.g., V600) must have failed or are intolerant to prior treatment with BRAF inhibitors

Inclusion Criteria Specific to Arm E (Atezolizumab +Obinutuzumab)

- R/M HNSCC participants with at least one prior line of systemic therapy

Inclusion Criteria Specific to prior Anti-PD-L1/PD-1 Treated Cohorts:

* No permanent discontinuation of atezolizumab or other immunotherapies due to a treatment-related adverse event
* Recovery from all immunotherapy-related adverse events to Grade less than or equal to (≤) 1 or baseline at the time of consent

Exclusion Criteria:

General Medical Exclusions:

* Pregnant and lactating women
* Any approved anti-cancer therapy, including chemotherapy or hormonal therapy, within 3 weeks prior to initiation of study treatment, with the following exception: (1) hormone-replacement therapy or oral contraceptives; (2) tyrosine kinase inhibitors (TKIs) that have been discontinued greater than (>) 7 days prior to Cycle 1, Day 1, baseline scans must be obtained after discontinuation of prior TKIs
* Investigational therapy within 28 days prior to initiation of study treatment
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity or allergy to Chinese hamster ovary cell products or any component of the atezolizumab formulation
* History of or active autoimmune disease
* History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia, risk of pulmonary toxicity, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Prior allogeneic bone marrow transplantation or prior solid organ transplantation
* History of human immunodeficiency virus (HIV)
* Participants with active hepatitis B
* Participants with active hepatitis C
* Participants with active tuberculosis
* Participants with a history of confirmed progressive multifocal leukoencephalopathy
* Any serious medical condition, physical examination finding, or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the participant's safe participation in and completion of the study

Cancer-Specific Exclusions:

* Active or untreated central nervous system (CNS) metastases, as determined by CT or magnetic resonance imaging (MRI) evaluation during screening and prior radiographic assessments
* Spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for >/= 2 weeks prior to screening
* Leptomeningeal disease
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently); participants with indwelling catheters are allowed.
* Uncontrolled tumor-related pain
* Uncontrolled hypercalcemia or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy or denosumab
* History of other malignancy within 2 years prior to screening, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, Stage I uterine cancer, localized prostate cancer treated with curative intent, ductal carcinoma in situ treated surgically with curative intent, or other cancers with a similar outcome

Exclusion Criteria Related to Medications:

* Prior treatment with cluster of differentiation 137 (CD137) agonists or immune checkpoint blockade therapies (Note: Participants enrolled in the prior anti-PD-L1/PD-1 treated cohorts with melanoma may have received prior anti-cytotoxic T-lymphocyte-associated protein 4 treatment or other immunotherapies)
* Treatment with systemic immunostimulatory agents within four weeks or five half-lives of the drug, whichever is shorter, prior to Cycle 1, Day 1
* Treatment with systemic immunosuppressive medications within 2 weeks prior to Cycle 1, Day 1 (the use of inhaled corticosteroids and mineralocorticoids is allowed)

Exclusion Criteria Specific to Interferon Alpha Therapy (Arms B-D):

* History of depression, suicidal ideation or behavior, bipolar disorder, or psychosis
* Hypersensitivity to interferon alpha or any component of the product

Exclusion Criteria Specific to Bevacizumab (Arm D)

* Inadequately controlled hypertension
* Prior history of hypertensive crisis or hypertensive encephalopathy
* Significant vascular disease within 6 months prior to Day 1
* History of hemoptysis
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* History of tracheoesophageal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 1
* Clinical signs or symptoms of gastrointestinal obstruction or requirement for routine parenteral hydration, parenteral nutrition, or tube feeding
* Evidence of abdominal free air that is not explained by paracentesis or recent surgical procedure
* Proteinuria, as demonstrated by urine dipstick or > 1.0 gram of protein in a 24-hour urine collection
* Metastatic disease that involves major airways or blood vessels, or centrally located mediastinal tumor masses of large volume

Exclusion Criteria Specific Obinutuzumab (Arm E)

* Hypersensitivity to obinutuzumab
* Prior treatment with obinutuzumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2014-08-18 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Recommended Phase II Dose (RP2D) of Atezolizumab When Given in Combination With Ipilimumab and Interferon Alfa-2b | From the first atezolizumab treatment up to 21 days
Percentage of Participants with Adverse Events | From the first atezolizumab treatment up to 4.5 years (yr)

SECONDARY OUTCOMES:
Percentage of Participants with Best Overall Response, as Assessed Using Conventional Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Screening to progression or death, up to 4.5 yr (assessed at baseline, every 6 weeks for 48 weeks and every 12 weeks thereafter up to treatment completion/early termination [up to 4.5 yr])
Percentage of Participants with Best Overall Response, as Assessed Using Immune Modified RECIST Criteria | Screening to progression or death, up to 4.5 years (assessed at baseline, every 6 weeks for 48 weeks and every 12 weeks thereafter up to treatment completion/early termination [up to 4.5 yr])
Duration of Objective Response | Screening to progression or death, up to 4.5 yr (assessed at baseline, every 6 weeks for 48 weeks and every 12 weeks thereafter up to treatment completion/early termination [up to 4.5 yr])
Overall Survival | Baseline to death (up to 4.5 yr)
Progression-Free Survival | Screening to progression or death, up to 4.5 yr (assessed at baseline, every 6 weeks for 48 weeks and every 12 weeks thereafter up to treatment completion/early termination [up to 4.5 yr])
Percentage of Participants with Objective Response, as Assessed Using Conventional RECIST v1.1 | Screening to progression or death, up to 4.5 yr (assessed at Baseline, every 6 weeks for 48 weeks and every 12 weeks thereafter up to treatment completion/early termination [up to 4.5 yr])
Percentage of Participants with Objective Response, as Assessed Using Immune Modified RECIST Criteria | Screening to progression or death, up to 4.5 yr (assessed at Baseline, every 6 weeks for 48 weeks and every 12 weeks thereafter up to treatment completion/early termination [up to 4.5 yr])
Serum Atezolizumab Concentration | Baseline up to 4.5 years (detailed timeframe is given in outcome description)
  Arm A: Predose (0 hour [hr]), 30 minutes (min) post end of infusion on Day 1;Day 8,Day 15 of Cycle (cy) 1;Predose (0 hr) on Day 1 of cy 2,3,4,8; end of treatment/withdrawal;≥ 90 days post last dose (up to 4.5 years [yr]). Arm B: Predose (0 hr) on Day 1,30 min post end of infusion on Day 8,Day 15,Day 22 of cy 1;Predose (0 hr) on Day 1 of cy 2,3,4,5,8; end of treatment/withdrawal;≥ 90 days post last dose (up to 4.5 yr). Arms C,D: Predose (0 hr), 30 min post end of infusion on Day 1 cy 1,3;Predose (0 hr) on Day 1 of cy 2,4,8, every 8 cy thereafter up to end of treatment/withdrawal;≥ 90 days post last dose (up to 4.5 yr). Arm E: Predose (0 hr), 30 min post end of infusion on Day 1 cy 1,5;Predose (0 hr) on Day 1 of cy 2,3,4,8, every 8 cy thereafter up to treatment end of treatment/withdrawal;≥ 90 days post last dose (up to 4.5 yr). Cycle length = 21 days (28 days for Arm B, cycle 1)
Serum Ipilimumab Concentration | Baseline up to 4.5 years (detailed timeframe is given in outcome description)
  Predose (0 hr), 30 min post end of infusion on Day 1 of Cy 1,3;Predose on Day 1 of Cy 4; end of treatment/ withdrawal;≥ 90 days post last dose (up to 4.5 yr) Cycle length = 21 days
Serum Bevacizumab Concentration | Baseline up to 4.5 years (detailed timeframe is given in outcome description)
  Predose (0 hr), 30 min post end of infusion on Day 1 of Cy 1,3; end of treatment/ withdrawal;≥ 90 days post last dose (up to 4.5 yr) Cycle length = 21 days
Serum Obinutuzumab Concentration | Baseline up to 4.5 years (detailed outcome given in outcome description)
  Predose (0 hr), 30 min post end of infusion on Days -13, -12 and on Day 1 Cy 5; end of treatment/withdrawal;≥90 days post last dose (up to 4.5 yr) Cycle length = 21 days
Anti-Drug Antibody to Atezolizumab | Baseline up to 4.5 years (detailed timeframe is given in outcome description)
  Detailed timeframe:
  Arm A: Predose (0 hr) on Day 1 of Cy 1,2,3,4,8; end of treatment/withdrawal;≥ 90 days post last dose (up to 4.5 yr).
  Arm B: Predose (0 hr) on Day 1 of Cy 1,2,3,4,5,8; end of treatment/withdrawal;≥ 90 days post last dose (up to 4.5 yr).
  Arms C, D, E: Predose (0 hr) on Day 1 of cy 1,2,3,4,8, thereafter every 8 Cy up to end of treatment/ withdrawal;≥ 90 days post last dose (up to 4.5 yr).
  Cycle length = 21 days (28 days for Arm B, cycle 1)
Anti-Drug Antibody to Ipilimumab | Baseline up to 4.5 years (detailed timeframe is given in outcome description)
  Pre-dose (0 hr) on Day 1 of Cy 1, 4, end of treatment/ withdrawal;≥ 90 days post last dose (up to 4.5 yr) Cycle length = 21 days
Anti-Drug Antibody to Bevacizumab | Baseline up to 4.5 years (detailed timeframe is given in outcome description)
  Predose (0 hr) on Day 1 of Cy 1, 3; end of treatment/withdrawal;≥ 90 days post last dose (up to 4.5 yr).
  Cycle length = 21 days
Anti-Drug Antibody to Obinutuzumab | Baseline up to 4.5 years (detailed timeframe is given in outcome description)
  Predose (0 hr) on Days -13 and -12; end of treatment/withdrawal;≥ 90 days post last dose (up to 4.5 yr) Cycle length = 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- United States (8):
  - HonorHealth Research Institute - Bisgrove, Scottsdale, Arizona
  - Mayo Clinic- Scottsdale, Scottsdale, Arizona
  - UCLA, Los Angeles, California
  - Yale University, New Haven, Connecticut
  - Mayo Clinic-Jacksonville, Jacksonville, Florida
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Sarah Cannon Research Inst., Nashville, Tennessee
  - Vanderbilt Medical Center, Nashville, Tennessee
- The Netherlands Cancer Institute of Amsterdam, Amsterdam, Netherlands